CLINICAL TRIAL: NCT03965052
Title: Phase I Clinical Study, to Evaluate the Safety and Tolerability of the Ophthalmic Solution PRO-179 Compared With Travatan®, on the Ocular Surface of Clinically Healthy Subjects.
Brief Title: Safety and Tolerability of the Ophthalmic Solution PRO-179 Compared With Travatan®
Acronym: PRO-179/I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Sophia S.A de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOPH179-0818/I
Record Dates: First submitted 2019-05-23; First posted 2019-05-28 (Actual); Results first posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-11

CONDITIONS: Glaucoma
Keywords: Travoprost; ophthalmic solution; Prostaglandin Analogues; Antiglaucoma drugs; glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Travoprost; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: double blind, with randomization.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding will correspond to the principal investigator and coinvestigator. In addition, the statistical analysis will be carried out in a blinded manner for the final analysis. Blinding can not be guaranteed in the subject.
  The masking will be done through the secondary container. The primary packaging will not be masked by the morphological difference between them. The sponsor and the research center will have two teams blinded / not blinded.
  They will be identified by means of identical labels. Which, in accordance with current and applicable regulations, must contain at least:
  * Name, address and telephone number of the sponsor.
  * Pharmaceutical form and route of administration.
  * Lot Number.
  * Legend "Exclusively for clinical studies"
  * Date of Expiry.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRO-179 (Experimental): Dosage: 1 drop every 24 hours, at night, in both eyes.
  Interventions: Drug: PRO 179
- Travatan® (Active Comparator): Dosage: 1 drop every 24 hours, at night, in both eyes.
  Interventions: Drug: Travatan 0.004 % Ophthalmic Solution

INTERVENTIONS:
Drug: PRO 179 — * Generic name: Travoprost
  * Distinctive denomination: Bristrio® (PRO-179)
  * Active principles: Travoprost 0.004%.
  * Pharmaceutical form: Ophthalmic solution
  * Presentation: multi-dose dropper bottle, 2.5 milliliters.
  * Prepared by: Sophia Laboratories, S.A. of C.V.
  * Description of the solution: transparent solution, free of visible particles.
  * Description of container: White bottle with 5 milliliters capacity, made of low density polyethylene.
  Other Names: PRO-179; Bristrio®; Travoprost 0.004% ophthalmic solution
  Arms: PRO-179
Drug: Travatan 0.004 % Ophthalmic Solution — * Generic name: Travoprost
  * Distinctive denomination: Travatan®
  * Active ingredients: Travoprost 0.004%
  * Pharmaceutical form: Ophthalmic solution.
  * Presentation: multi-dose dropper bottle, 2.5 milliliters.
  * Prepared by: Alcon Laboratories Inc.
  * Description of the solution: transparent solution, free of visible particles.
  * Consult information to prescribe.
  Other Names: Travoprost 0.004% ophthalmic solution
  Arms: Travatan®

SUMMARY:
Phase I clinical study, to evaluate the safety and tolerability of the ophthalmic solution PRO-179 compared with Travatan®, on the ocular surface of clinically healthy subjects.

Goals: To evaluate the safety and tolerability of the formulation PRO-179 manufactured by Sophia Laboratories S.A. of C.V. on the ocular surface of clinically healthy subjects.

Hypothesis:The ophthalmic solution PRO-179 presents a profile of safety and tolerability similar to Travatan® in healthy subjects.

Methodology: Clinical trial Phase I, controlled, of parallel groups, double blind, with randomization.

DETAILED DESCRIPTION:
Number of patients: n= 24, 12 subjects per group (both eyes). Main inclusion criteria: Clinically healthy subjects.

duration: 10 days.

Duration of subject in the study: 15 to 22 days.

Adverse events will be reported and cataloged based on the MedDRA dictionary and will be reported to the corresponding regulatory entity.

The sponsor will carry out monitoring or quality visits to the research sites where it corroborates the information of the source documents and will contrast them with the information presented in the electronic CRF. Electronic case report forms will be evaluated by the clinical research associate and the clinical team of the sponsor (medical ophthalmologist researcher and pharmacologist of clinical safety).

Statistical methodology:

The data will be expressed with measures of central tendency: mean and standard deviation for the quantitative variables. The qualitative variables will be presented in frequencies and percentages. The statistical analysis will be carried out by means of the Mann-Whitney U test for the quantitative variables for the difference between the groups. The difference between the qualitative variables will be analyzed by means of X2 (Chi2) or Fisher's exact. An alpha ≤ 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Be clinically healthy.
* Have the ability to give their signed informed consent and show willingness to comply with the study procedures
* Have an age between 18 to 45 years.
* Indistinct sex.
* Women should ensure the continued use of a hormonal contraceptive method or intrauterine device (IUD) during the study period.
* Present blood tests: within normal parameters or with a range of ± 20% as long as the subject is clinically healthy.

Blood count (BH): Hemoglobin, erythrocytes, hematocrit, total leukocytes, platelets, mean corpuscular volume and mean corpuscular hemoglobin.

* Blood chemistry of three elements (QS): Glucose, urea and creatinine.
* Liver function tests (PFH): Aspartate Aminotransferase and Alanine Aminotransferase, total bilirubin, direct and indirect.

  * Present visual ability 20/30 or better in both eyes.
  * Present vital signs within normal parameters.
  * Present intraocular pressure ≥10 and ≤ 21 mmHg.

Exclusion Criteria:

* Be a user of topical ophthalmic products of any kind.
* Be a user of medicines, or herbal products, by any other route of administration, with the exception of hormonal contraceptives in the case of women.
* In case of being a woman, being pregnant or breastfeeding.
* Have participated in clinical research studies 90 days prior to inclusion in the present study.
* Have previously participated in this same study.
* Be a user of contact lenses and can not suspend their use during the study.
* That they can not follow the lifestyle considerations described in section 6.2.2
* Having started the use of hormonal contraceptives or IUD, 30 days prior to inclusion in the present study.
* Having a history of any chronic-degenerative disease.
* Present inflammatory or infectious disease, active at the time of admission to the study.
* Present injuries or unresolved traumas at the time of entering the study.
* Having the antecedent of any type of eye surgery.
* Having undergone surgical procedures, not ophthalmological, in the last 3 months.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Baiza Durán, MD, Study Director — Laboratorios Sophia S.A de C.V.
Locations (1):
- Jose Navarro Partida, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Munoz-Villegas P, Navarro-Sanchez AA, Sanchez-Rios A, Olvera-Montano O, Baiza-Duran LM. Reexamining Ophthalmic Drugs, Safety and Tolerability in Phase 1 Clinical Trials. Ther Clin Risk Manag. 2021 Oct 21;17:1123-1134. doi: 10.2147/TCRM.S331294. eCollection 2021. PMID 34707360

RESULTS

PARTICIPANT FLOW:
Groups:
- PRO-179: Dosage: 1 drop every 24 hours, at night, in both eyes.
  PRO 179: o Generic name: Travoprost
  * Distinctive denomination: Bristrio® (PRO-179)
  * Active principles: Travoprost 0.004%.
  * Pharmaceutical form: Ophthalmic solution
  * Presentation: multi-dose dropper bottle, 2.5 milliliters.
  * Prepared by: Sophia Laboratories, S.A. of C.V.
  * Description of the solution: transparent solution, free of visible particles.
  * Description of container: White bottle with 5 milliliters capacity, made of low density polyethylene.
- Travatan®: Dosage: 1 drop every 24 hours, at night, in both eyes.
  Travatan 0.004 % Ophthalmic Solution: o Generic name: Travoprost
  * Distinctive denomination: Travatan®
  * Active ingredients: Travoprost 0.004%
  * Pharmaceutical form: Ophthalmic solution.
  * Presentation: multi-dose dropper bottle, 2.5 milliliters.
  * Prepared by: Alcon Laboratories Inc.
  * Description of the solution: transparent solution, free of visible particles.
  * Consult information to prescribe.
Period: Overall Study
Arm/Group | PRO-179 | Travatan®
Started | 12 | 12
Completed | 11 | 12
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRO-179 | Travatan® | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (8.0) | 24.7 (4.6) | 26.3 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 8 | 4 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Latin | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  Mexico | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: primary security variable the adverse events will be evaluated with a scale of Present / Absent, it is a nominal variable, the normal value is absent. it will be evaluated by the number of reported cases per group.
Time Frame: during the 14 days of evaluation, including the safety call (day 14).
Population: the analysis was carried out by intention to treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | PRO-179 | Travatan®
Number analyzed (Participants) | 12 | 12
Participants | 10 | 11
Statistical Analysis 1: Comparison: PRO-179 vs Travatan®; Test type: Other; p = 1.000, Fisher Exact

2. Primary Outcome: Eye Comfort Index
Description: It is a questionnaire designed to measure the irritation of the ocular surface with Rasch analysis to produce estimates on a linear scale of intervals (ratings: 0-100).The Eye comfort index contains items that focus on the discomfort associated with alterations of the ocular surface.(0: None discomfort, 100: high discomfort).
Time Frame: will be evaluated at the end of the treatment, at the final visit (day 11)
Population: the analysis was per protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PRO-179 | Travatan®
Number analyzed (Participants) | 11 | 12
score on a scale | 26.61 (11.3) | 28.97 (7.9)

3. Secondary Outcome: Number of Eyes With Epithelial Defects by Grade
Description: The epithelial defects will be evaluated by means of two stains, lissamine green and fluorescein, it is a discrete variable that will be realized by direct observation, it will be staged according to the degrees of the oxford scale that go from 0 to 5 (0-V) according to its severity, where 0 is the normal lower limit and 5 the upper limit of defects.
Time Frame: will be evaluated at the end of the treatment, at the final visit (day 11)
Population: The analysis was per protocol
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-179 | Travatan®
Number analyzed (Participants) | 11 | 12
Number analyzed (eyes) | 22 | 24
eyes
  Green lissamine grade 0 | 22 | 23
  Green lissamine grade 1 | 0 | 1
  Green lissamine grade 2 | 0 | 0
  Green lissamine grade 3 | 0 | 0
  Green lissamine grade 4 | 0 | 0
  Fluorescein grade 0 | 20 | 20
  Fluorescein grade 1 | 2 | 4
  Fluorescein grade 2 | 0 | 0
  Fluorescein grade 3 | 0 | 0
  Fluorescein grade 4 | 0 | 0
Statistical Analysis 1: Comparison: PRO-179 vs Travatan®; Lissamine green treatment groups; Test type: Other; p = 1.000, Fisher Exact
Statistical Analysis 2: Comparison: PRO-179 vs Travatan®; Fluorescein treatment groups; Test type: Other; p = 0.667, Fisher Exact

4. Secondary Outcome: Visual Ability
Description: The visual capacity variable will be reported using as a unit of measure a fraction, this is taken from a visual test with the Snellen primer, it is a Nominal type variable. where the optimal vision is 20/20 and the worst vision is 20/200, higher values represent a worst vision. The result of the Snellen chart has equivalents in an international logarithmic system called Logmar (logarithm of the minimum angle of resolution) for better understanding.
  Snellen Scale: 20/200, 20/100, 20/50, 20/40, 20/30, 20/25, 20/20, 20/15, 20/12, 20/10.
  Snellen / LogMAR equivalences: 20/200= 1.0, 20/100=0.7, 20/50=0.4, 20/40=0.3, 20/30=0.2, 20/25=0.1, 20/20=0.0, 20/15=0.13, 20/12=0.2, 20/10=-0.3, etc.
Time Frame: will be evaluated at the end of the treatment, at the final visit (day 11)
Population: the analysis was per protocol
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | PRO-179 | Travatan®
Number analyzed (Participants) | 11 | 12
LogMAR | 0.0 (0) | 0.0 (0)
Statistical Analysis 1: Comparison: PRO-179 vs Travatan®; Test type: Other; p = 1.000, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Percentage of Eyes With Conjunctival Hyperemia (CH) by Grade
Description: Conjunctival hyperemia will be evaluated as an ordinal variable, by direct observation and staged using the Efron scale as Normal / Very Light / Mild / Moderate / Severe. Based on this scale, the normal and mild stages are considered without pathologies or normal. Mild, moderate and severe are considered pathological.
Time Frame: will be evaluated at the end of the treatment, at the final visit (day 11)
Population: the analysis was per protocol
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-179 | Travatan®
Number analyzed (Participants) | 11 | 12
Number analyzed (eyes) | 22 | 24
eyes
  Normal (0) | 14 | 16
  Very mild (1) | 2 | 2
  Mild (2) | 6 | 6
  Moderate (3) | 0 | 0
  Severe (4) | 0 | 0
Statistical Analysis 1: Comparison: PRO-179 vs Travatan®; the analysis was per protocol; Test type: Other; p = 0.977, Chi-squared, Corrected

6. Secondary Outcome: Number of Eyes of Chemosis
Description: The chemosis will be evaluated, as a nominal variable, by direct observation and it will be staged as present and absent, where the normality is that said variable is absent.
Time Frame: will be evaluated at the end of the treatment, at the final visit (day 11)
Population: the analysis was per protocol
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | PRO-179 | Travatan®
Number analyzed (Participants) | 11 | 12
Number analyzed (eyes) | 22 | 24
eyes | 0 | 0

7. Other Pre Specified Outcome: Changes in Intraocular Pressure
Description: the intraocular pressure will be evaluated by means of the Goldman applanation tonometry whose unit of measurement is millimeters of mercury (mmHg), it is a continuous variable and its normality range is between 11 - 21 mmHg
Time Frame: will be evaluated at the end of the treatment, at the final visit (day 11)
Population: the analysis was per protocol
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: eyes
Arm/Group | PRO-179 | Travatan®
Number analyzed (Participants) | 11 | 12
Number analyzed (eyes) | 22 | 24
mmHg | 11.95 (1.6) | 10.71 (1.5)
Statistical Analysis 1: Comparison: PRO-179 vs Travatan®; Test type: Other; p = 0.019, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Adverse events were evaluated for about 2 months and one week until the last follow-up call of the last subject.
Arm/Group | PRO-179 | Travatan®
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/12
Other Adverse Events (participants affected / at risk) | 10/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-179 (N=12) | Travatan® (N=12)
ocular hypotony (Eye disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRO-179 (N=12) | Travatan® (N=12)
ocular burning (Eye disorders) | 4 (4) | 6 (6)
headache (Nervous system disorders) | 0 (0) | 1 (1)
eye pain (Eye disorders) | 2 (2) | 2 (2)
eyelid pain (Eye disorders) | 0 (0) | 1 (1)
photophobia (Eye disorders) | 2 (2) | 1 (1)
ocular hypotony (Eye disorders) | 1 (1) | 1 (1)
eyelid swelling (Eye disorders) | 1 (1) | 1 (1)
tearing (Eye disorders) | 0 (0) | 2 (2)
red eye (Eye disorders) | 10 (10) | 9 (9)
eye itching (Eye disorders) | 2 (2) | 3 (3)
Eye discharge (Eye disorders) | 1 (1) | 0 (0)
foreign body sensation (Eye disorders) | 0 (0) | 1 (1)
Dry eye (General disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator undertakes not to publish or communicate data collected from the study, unless there is prior written agreement of Laboratorios Sophia, S.A. from C.V.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT03965052/Prot_SAP_000.pdf